CLINICAL TRIAL: NCT02924597
Title: Robot-Assisted Laparoscopic Radio Frequency Ablation Assisted Enucleation of Renal Cell Carcinoma With T1a Stage : Clinical Outcomes of a Randomised Controlled Trial
Brief Title: Robot-Assisted Laparoscopic Radio Frequency Ablation Assisted Enucleation of Renal Cell Carcinoma With T1a Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RenJiH-20160829
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted laparoscopic RFA assisted TE (Experimental): RFA will be performed for 1 to 4 cycles for 4 to 12 minutes each depending on tumor size and depth. The tumor then will be laparoscopic enucleation without hilar clamping.
  Interventions: Procedure: zero ischemia robot-assisted laparoscopic RFA assisted TE
- Robot-Assisted laparoscopic partial nephrectomy (Active Comparator): The tumor then will be laparoscopic enucleation without hilar clamping.
  Interventions: Procedure: zero ischemia robot-assisted laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: zero ischemia robot-assisted laparoscopic RFA assisted TE
  Other Names: zero ischemia robot-assisted laparoscopic radio frequency ablation assisted tumor enucleation
  Arms: Robot-assisted laparoscopic RFA assisted TE
Procedure: zero ischemia robot-assisted laparoscopic partial nephrectomy
  Other Names: Off-clamp robot-assisted partial nephrectomy
  Arms: Robot-Assisted laparoscopic partial nephrectomy

SUMMARY:
To evaluate the feasibility and efﬁciency of zero ischemia robot-assisted laparoscopic radio frequency ablation assisted enucleation of T1a renal cell carcinoma in comparison with robot-assisted laparoscopic partial nephrectomy without hilar clamping.

ELIGIBILITY:
Inclusion Criteria:

* patients with sporadic, unilateral, newly diagnosed T1a presumed renal cell carcinoma
* patients scheduled for robot-assisted laparoscopic nephron sparing surgery
* patients with normal contralateral renal function (diﬀerential renal function of >40% as determined by radionuclide scintigraphy)
* patients agreeable to participate in this long-term follow-up study

Exclusion Criteria:

* patients' aged >80 years
* patients with other renal diseases,(including kidney stone, glomerular nephritis, etc.) which might affect the renal function of the operative kidney
* patients not able to tolerate the robot-assisted laparoscopic procedure
* patients with previous renal surgery or history of any inﬂammatory conditions of the operative kidney
* patients with the renal tumor involving urinary collecting system

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The absolute change in glomerular ﬁltration rate (GFR) of the aﬀected kidney | baseline and 12 months
  12 months minus baseline
The changes of estimated GFR (eGFR) | baseline and 12 months
  12 months minus baseline

SECONDARY OUTCOMES:
estimated blood loss | during surgery
changes in GFR of total kidneys by renal scintigraphyby | baseline and 12 months
surgical margin | postoperative，up to 2 weeks after surgery
postoperative complications | postoperative，up to 30 days
progression-free survival | 12 months
local recurrence | 12 months
operative time | During surgery
Hospital stay time | The time from the surgery day to patient discharge, up to 2 weeks
changes in GFR of total kidneys by renal scintigraphyby of 6 month | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China